CLINICAL TRIAL: NCT00040469
Title: Allogeneic Bone Marrow Transplant From HLA Identical Related Donors for Patients With High Risk Hemoglobinopathies: Hemoglobin SS, Hemoglobin SC, Hemoglobin SB0/+ Thalassemia, or Homozygous B0/+ Thalassemia or Severe Variants of B0/+ Thalassemia
Brief Title: Bone Marrow Transplant From Related Donor for Patients With High Risk Hemoglobinopathies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual was slow and sporadic so the study was closed
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H6847; Scallo2
Record Dates: First submitted 2002-06-26; First posted 2002-06-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Anemia; Hemoglobinopathy; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Thalassemia | interventions — Alemtuzumab; Phenytoin; Busulfan; Cyclophosphamide

INTERVENTIONS:
Drug: Campath -1H
Drug: Dilantin
Drug: Busulfan
Drug: Cyclophosphamide

SUMMARY:
The major goal of this study is to determine the risks and benefits of bone marrow transplants in patients with severe thalassemia or sickle cell disease. Participation in this project will be for two years.

DETAILED DESCRIPTION:
To do the bone marrow transplant, we must first kill the cells in the bone marrow that make the abnormal red blood cells that are found in patients with severe thalassemia or sickle cell disease.

We will do this by using three drugs: busulfan, cyclophosphamide, and CAMPATH-1H. CAMPATH-IH is an investigational drug. CAMPATH-1H is used to prevent participants from rejecting or refusing to let the donor blood cells grow in the body. After the drug treatment, participants will be given bone marrow from a brother or sister who has healthy bone marrow that matches.

ELIGIBILITY:
Inclusion:

* Patients with homozygous B0/+ thalassemia or severe variants of B0/+ thalassemia with an HLA genotypically identical donor.
* Patients with an HLA genotype identical donor and hemoglobin SS, hemoglobin SC, or hemoglobin Sb 0/+ and at least one of the following:

Previous central nervous system vaso-occlusive episode with or without residual neurologic findings; Frequent painful vaso-occlusive episodes which significantly interfere with normal life activities and which necessitate chronic transfusion therapy; Recurrent SCD chest syndrome events which necessitate chronic transfusion therapy.

* Severe anemia which prevents acceptable quality of life and necessitates chronic transfusion therapy.
* The patient must have an HLA genotype identical donor.
* Between the ages of birth and 65 years.
* Women of childbearing potential must have a negative pregnancy test.

Exclusion:

* Biopsy proven chronic active hepatitis or fibrosis with portal bridging.
* SCD chronic lung disease >/= stage 3.
* Severe renal dysfunction defined as creatinine clearance <40 ml/min/1.73 M2
* Severe cardiac dysfunction defined as shortening fraction <25%.
* HIV infection.
* Severe but unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplant (BMT).
* Inadequate intellectual capacity to understand the nature and risk inherent in the BMT process and give informed consent (in the case of minors, this criteria must be fulfilled by the legal guardian).
* Pregnant, lactating or unwilling to use appropriate birth control.

Ages: 1 Day to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15
Dates: Start 2000-08; Primary Completion 2003-11-21 (Actual); Study Completion 2003-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K. Brenner, MD, Study Chair — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas